CLINICAL TRIAL: NCT06389370
Title: Assessment of Oral Health Knowledge, Attitude and Behaviour and Its Association With Sociodemographic Factors of Preclinical and Clinical Dental Students in Cairo University: A Cross-Sectional Study
Brief Title: Assessment of Oral Health Knowledge, Attitude and Behaviour of Dental Students in Cairo University
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alyaa Ibrahim Abbas Ahmed, principle investigator, Cairo University
Other Study IDs: knowledge, Attitude, Behaviour
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Oral Health Knowledge, Attitude and Behaviour of Dental Students
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Level 1
  Interventions: Other: HU-DBI questionnaire
- Level 2
  Interventions: Other: HU-DBI questionnaire
- Level 3
  Interventions: Other: HU-DBI questionnaire
- Level 4
  Interventions: Other: HU-DBI questionnaire
- Level 5
  Interventions: Other: HU-DBI questionnaire

INTERVENTIONS:
Other: HU-DBI questionnaire — a questionnaire published by Hiroshima University (HU-DBI) to measure the Knowledge, Attitude and Behaviour of dental students through different levels of their academic years.

SUMMARY:
The knowledge, behaviour and attitude of oral health professionals reflects their awareness and understanding of oral preventive measures, which will have significant impact on their delivery of public oral health promotion in the future. They are expected to set an example for positive oral health behaviour among other college students, family members and their patients. Various external factors like sociodemographic factors like age, gender, marital state, occupation, and number of family members play a major role in oral hygiene. The relationships between various modifiable factors needs to be assesses in a vast manner.

There were some researches about oral health knowledge, behaviour and attitude in correlation to socio-demographic data, of dental students in other countries, but little was known in Egypt. Dental students are expected to play a critical role in instructing public oral health for improving their patient's, families, and friends. In addition, it may pave the way to develop new programs to encourage needful oral health practices.

ELIGIBILITY:
Inclusion Criteria:

* Preclinical and clinical dental students, Faculty of Dentistry, Cairo University through the academic year 2024-2025.

Exclusion Criteria:

* Dental students from other universities.
* Internship dental students.
* Post-graduate dental students.

Ages: 17 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Dental Students from level 1 to level 5 in faculty of dentistry, Cairo university.
Sampling Method: Probability Sample
Enrollment: 535 (Estimated)
Dates: Start 2024-11-04 (Estimated); Primary Completion 2024-11-18 (Estimated); Study Completion 2024-12-03 (Estimated)

PRIMARY OUTCOMES:
Knowledge | 1 month
  Items no. in the questionnaire: 2,8,10,15,19 will be measured dichotomous (Agree/Disagree) with minimum score 0 and maximum score 12

SECONDARY OUTCOMES:
Attitude and behaviour | 1 month
  Attitude will be items no. 6,11,14 and Behviour will be items 4,9,12,16 will be measured dichotomous (Agree/Disagree) with minimum score 0 and maximum score 12

CONTACTS AND LOCATIONS:
Overall Officials: Alyaa IA Ahmed, BDS, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided
Data to be shared is the results of KAB scores and the statistics of these results.